CLINICAL TRIAL: NCT00282984
Title: A 12-Week, Double-Blind, Placebo-Controlled, Multicenter Study With A 40 Week Follow Up Evaluating the Safety and Efficacy of Varenicline Tartrate 1 Milligram (Mg) Twice Daily (BID) for Smoking Cessation in Subjects With Cardiovascular Disease
Brief Title: Efficacy and Safety of Varenicline in Smokers With Cardiovascular Disease Who Wish to Quit Smoking
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3051049
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2009-04-29 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- varenicline (Experimental)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: placebo — 1 mg placebo twice daily by mouth for 12 weeks
  Arms: placebo
Drug: Varenicline — 1 mg twice daily by mouth for 12 weeks
  Other Names: Chantix, Champix
  Arms: varenicline

SUMMARY:
The primary purpose of this study is to determine whether or not varenicline will help people with cardiovascular disease quit smoking and to confirm it is safe in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have stable, documented cardiovascular disease (including at least one of the following diagnosed > 2 months prior to the Screening visit - angina, myocardial infarction (MI), revascularization, transient ischemic attack (TIA), and peripheral vascular disease (PVD).
* Participants that smoke > 10 cigarettes / day.

Exclusion Criteria:

* Participants with unstable cardiovascular disease
* Cardiovascular events in the past 2 months
* Moderate or severe chronic obstructive pulmonary disease (COPD)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2006-02; Primary Completion 2007-11 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (3):
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Madison, Wisconsin
- Argentina (2):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, Ciudad de Buenos Aires, Buenos Aires
- Australia (2):
  - Pfizer Investigational Site, Concord, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (4):
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Drummondville, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Czechia (2):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
- Denmark (2):
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Hellerup
- France (3):
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Toulouse
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Tübingen
- Greece (2):
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Pireaus
- Mexico (2):
  - Pfizer Investigational Site, Tlalpan, Mexico City
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Netherlands (2):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Zuthpen
- South Korea (2):
  - Pfizer Investigational Site, Seoul, Korea
  - Pfizer Investigational Site, Seoul
- Taiwan (2):
  - Pfizer Investigational Site, Taipei, Taiwan
  - Pfizer Investigational Site, Tau-Yuan Hsien
- United Kingdom (4):
  - Pfizer Investigational Site, Carshalton, Surrey
  - Pfizer Investigational Site, Bradford, West Yorkshire
  - Pfizer Investigational Site, Leicester
  - Pfizer Investigational Site, Paisley

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Rigotti NA, Pipe AL, Benowitz NL, Arteaga C, Garza D, Tonstad S. Efficacy and safety of varenicline for smoking cessation in patients with cardiovascular disease: a randomized trial. Circulation. 2010 Jan 19;121(2):221-9. doi: 10.1161/CIRCULATIONAHA.109.869008. Epub 2010 Jan 4. PMID 20048210
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051049&StudyName=Effectiveness%20and%20Safety%20of%20Varenicline%20in%20Smokers%20with%20Cardiovascular%20Disease%20Who%20Wish%20to%20Quit%20Smoking

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in outpatients. The target population was cigarette smokers with cardiovascular disease drawn from the communities surrounding the participating clinics.
Pre-assignment Details: 714 smokers were randomized (ie, assigned to study treatment), 11 participants were randomized, but not treated. The reasons for participants being randomized, not treated included no longer willing to participate in the study (5 participants), protocol violation (3 participants), lost to follow-up (1 participant), and other (2 participants).
Groups:
- Varenicline (Var): 1 week titration followed by 11 weeks of 1 milligram (mg) twice daily (BID) dosing. Study medication was discontinued at the Week 12 visit and participants' smoking status was followed through the non-treatment period to Week 52.
- Placebo (Pbo): 1 week titration followed by 11 weeks of placebo (pbo). Study medication was discontinued at the Week 12 visit and participants' smoking status was followed through the non-treatment period to Week 52.
Period: Overall Study
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Started | 353 | 350
Completed | 302 | 289
Not Completed | 51 | 61
Not completed — Death | 2 | 5
Not completed — Adverse Event | 8 | 5
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 14 | 10
Not completed — Withdrawal by Participant | 22 | 34
Not completed — Participant stopped study medication | 2 | 2
Not completed — Participant only allowed phone follow-up | 0 | 1
Not completed — Participant used antipsychosis meds | 0 | 1
Not completed — lack of motivation | 1 | 0
Not completed — in prison | 0 | 1
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline (Var) | Placebo (Pbo) | Total
Number analyzed (Participants) | 353 | 350 | 703
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (8.6) | 56.0 (8.4) | 56.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 63 | 150
  Male | 266 | 287 | 553

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders With Carbon Monoxide (CO) Confirmed 4-week Continuous Quit Rate (CQR) for Last 4 Weeks of Treatment (Trtmt)
Description: Participants considered Responders (4-week CQR <=10 parts per million <ppm>) through reports of cigarette or other nicotine use since last study visit, confirmed by measurement of end-expiratory exhaled carbon monoxide (CO). If any CO measurement at a particular timepoint was >10 ppm, subject was considered to be Non-Responder at that timepoint.
Time Frame: weeks 9 through 12
Population: Primary analysis population (Modified Intent-to-Treat) included all participants who took at least 1 dose randomized study medication. Participants who discontinued study were assumed smokers from timepoint of discontinuation through end of study. Modified Intent-to-Treat population is referred to as "All Participants" population in this report.
Measure: Number; unit: participants
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
participants
  responders | 167 | 50
  non-responders | 186 | 300
Statistical Analysis 1: Comparison: Varenicline (Var) vs Placebo (Pbo); Estimates for expected & clinically meaningful var & pbo 4-week CQR for Week 9 - 12 of trtmt based on response rates & corresponding 95% OR confidence interval (CI) from A30510285 & A30510366 study results. Total n=700 randomized var or pbo 1:1 should have provided at least 99% power to detect difference in primary endpoint (endpt) between (b/w) var & pbo, assuming true 4-week CQR of 0.18 for pbo & 0.40 for var (OR of at least 3.04), and 84% power for 2 key secondary endpts; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — To preserve type I family-wise error rate of 0.05, used step-down procedure to analyze primary & 2 key secondary endpoints. Hierarchy of comparisons: 1) 4-week CQR for Weeks 9 thru 12, 2) CA at Week 52, 3) the Long Term Quit Rate (LTQR) thru Week 52; Logistic regression model fitted to primary endpoint & key secondary endpoints; included main effects of trtmt group and center as independent var; Odds Ratio (OR) = 6.05, 95% CI [4.13 to 8.86]

2. Secondary Outcome: Number of Responders With Continuous Abstinence (CA) Through Week 52
Description: Responders: participants who remained abstinent based on 'since the last contact' question in Nicotine Use Inventory 1) "Has participant smoked any cigarettes (even a puff) since last contact?" = No AND 2) "Has participant used any other tobacco products… since last contact?" = No. Participant a non-responder if expired CO > 10 ppm.
Time Frame: Week 9 through Week 52
Population: All participants population
Measure: Number; unit: participants
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
participants
  responders | 70 | 26
  non-responders | 283 | 324
Statistical Analysis 1: Comparison: Varenicline (Var) vs Placebo (Pbo); Estimates for expected and clinically meaningful var & pbo 4-week CQR for Weeks 9 - 12 of trtmt were based on response rates & corresponding 95% odds ratio CI from A30510285 and A30510366 study results. Total n=700 randomized var or pbo 1:1 should have provided at least 99% power to detect difference in primary endpt b/w var & pbo, assuming true 4-week CQR of 0.18 for pbo & 0.40 for var (odds ratio of at least 3.04) & a power of 84% for the 2 key secondary endpts; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — To preserve type I family-wise error rate of 0.05, a step-down procedure was used for the analysis of primary & 2 key secondary endpts. Hierarchy of comparisons: 1) 4-week CQR for Weeks 9 through 12, 2) CA at Week 52, 3) LTQR through Week 52; Logistic regression model fitted to primary endpoint & key secondary endpoints; included main effects of treatment group & center as independent var; Odds Ratio (OR) = 3.19, 95% CI [1.97 to 5.18]

3. Secondary Outcome: Number of Long-Term Quit Responders
Description: Responders: participants were considered Long Term Quit responders if 1) they were responders for the primary endpoint (the 4-week CQR for Weeks 9-12) and 2) had no more than 6 days of smoking from Week 12 through the given visit.
Time Frame: Week 9 through Week 52
Population: All participants population
Measure: Number; unit: participants
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
participants
  responders | 80 | 34
  non-responders | 273 | 316
Statistical Analysis 1: Comparison: Varenicline (Var) vs Placebo (Pbo); Estimates for expected and clinically meaningful varenicline (var) & pbo 4-week CQR for Weeks 9 - 12 of treatment were based on response rates & corresponding 95% odds ratio CI from A30510285 and A30510366 study results. Total n=700 randomized var or pbo 1:1 should have provided at least 99% power to detect difference in primary endpt b/w varenicline & pbo, assuming true 4-week CQR of 0.18 for pbo & 0.40 for var (odds ratio of at least 3.04), and a power of 84% for the 2 key secondary endpts; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — To preserve type I family-wise error rate of 0.05, a step-down procedure was used for the analysis of primary & 2 key secondary endpoints. Hierarchy of comparisons: 1) 4-week CQR for Weeks 9 through 12, 2) CA at Week 52, 3) the LTQR through Week 52; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.82, 95% CI [1.82 to 4.38]

4. Secondary Outcome: Number of Participants With a Seven-Day Point Prevalence of Abstinence at Week 12
Description: Responders: abstinence in previous seven days, defined in the non-treatment follow-up as: 1) "Has the participant smoked any cigarettes in the last 7 days?" = No AND 2) "Has the participant used any other tobacco products in the last 7 days?" = No. Participant a non-responder if expired CO > 10 ppm.
Time Frame: Week 12
Population: All Participants population
Measure: Number; unit: participants
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
participants
  responders | 192 | 65
  non-responders | 161 | 285
Statistical Analysis 1: Comparison: Varenicline (Var) vs Placebo (Pbo); Week 12 analysis; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.97, 95% CI [4.17 to 8.56]

5. Secondary Outcome: Number of Participants With a Seven-Day Point Prevalence of Abstinence at Week 24
Description: as for outcome 4
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
participants
  responders | 124 | 57
  non-responders | 229 | 293
Statistical Analysis 1: Comparison: Varenicline (Var) vs Placebo (Pbo); 24 Week analysis; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.93, 95% CI [2.03 to 4.23]

6. Secondary Outcome: Number of Participants With a Seven-Day Point Prevalence of Abstinence at Week 52
Description: as for outcome 4
Time Frame: Week 52
Measure: Number; unit: participants
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
participants
  responders | 102 | 62
  non-responders | 251 | 288
Statistical Analysis 1: Comparison: Varenicline (Var) vs Placebo (Pbo); 52 Week analysis; Test type: Superiority or Other; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 1.93, 95% CI [1.34 to 2.77]

7. Secondary Outcome: Number of Participants With a 4 Week Point Prevalence of Smoking Cessation
Description: Responders: participants with abstinence during the last 4 weeks of non-treatment based on answering 'no' to both of the two 'last 4 week' questions in the Nicotine Use Inventory (NUI). NUI collected information of cigarette or other nicotine use during the study.
Time Frame: Week 48 through Week 52 (final 4 weeks of non-treatment period [pd])
Population: All Participants population
Measure: Number; unit: participants
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
participants | 99 | 57
Statistical Analysis 1: Comparison: Varenicline (Var) vs Placebo (Pbo); Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.05, 95% CI [1.41 to 2.97]

8. Secondary Outcome: Number of Responders With Continuous Abstinence (CA) Through Week 24
Description: Responders: participants who remained abstinent based on 'since the last contact' question in Nicotine Use Inventory 1) "Has participant smoked any cigarettes (even a puff) since the last contact?" = No AND 2) "Has participant used any other tobacco products… since the last contact?" = No. Non- responder if the expired CO > 10 ppm at any given timepoint.
Time Frame: Week 9 through Week 24
Population: All Participants population
Measure: Number; unit: participants
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
participants | 100 | 34
Statistical Analysis 1: Comparison: Varenicline (Var) vs Placebo (Pbo); Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.86, 95% CI [2.51 to 5.93]

9. Secondary Outcome: Cigarettes Smoked Per Day
Description: Cigarettes smoked each day during the first 3 weeks of the treatment phase.
Time Frame: Day 21
Population: All Participants population
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
cigarettes per day
  Baseline | 22.2 (10.0) | 22.9 (10.9)
  Day 1 | 17.6 (9.4) | 19.1 (10.0)
  Day 2 | 16.8 (8.8) | 18.4 (9.6)
  Day 3 | 15.8 (9.2) | 18.0 (10.0)
  Day 4 | 15.7 (8.9) | 17.1 (9.6)
  Day 5 | 15.1 (8.8) | 16.3 (8.9)
  Day 6 | 14.4 (8.4) | 16.0 (8.9)
  Day 7 | 13.8 (8.6) | 15.1 (8.8)
  Day 8 | 11.7 (9.2) | 12.3 (10.5)
  Day 9 | 9.5 (7.5) | 10.9 (9.5)
  Day 10 | 8.9 (7.2) | 10.6 (8.6)
  Day 11 | 8.9 (7.3) | 10.4 (8.4)
  Day 12 | 8.7 (7.5) | 10.5 (8.3)
  Day 13 | 8.8 (7.1) | 10.3 (8.2)
  Day 14 | 9.3 (7.4) | 10.7 (8.6)
  Day 15 | 8.9 (7.6) | 11.2 (9.1)
  Day 16 | 8.8 (7.1) | 11.0 (8.7)
  Day 17 | 8.3 (6.4) | 10.6 (8.2)
  Day 18 | 8.2 (6.9) | 10.3 (8.8)
  Day 19 | 7.8 (6.7) | 10.3 (8.4)
  Day 20 | 7.9 (6.1) | 10.6 (8.3)
  Day 21 | 7.2 (6.3) | 9.3 (8.1)

10. Secondary Outcome: Number of Long-Term Quit Responders From Week 9 Through Week 24
Description: as for outcome 3
Time Frame: Week 9 through Week 24
Population: All Participants population
Measure: Number; unit: participants
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Number analyzed (Participants) | 353 | 350
participants
  responders | 117 | 42
  non-responders | 236 | 308
Statistical Analysis 1: Comparison: Varenicline (Var) vs Placebo (Pbo); Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.85, 95% CI [2.58 to 5.75]

ADVERSE EVENTS:
Arm/Group | Varenicline (Var) | Placebo (Pbo)
Serious Adverse Events (participants affected / at risk) | 23 | 21
Other Adverse Events (participants affected / at risk) | 253 | 179
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Varenicline (Var) | Placebo (Pbo)
Anaemia (Blood and lymphatic system disorders) | 0/353 | 1/350
Acute coronary syndrome (Cardiac disorders) | 0/353 | 1/350
Acute myocardial infarction (Cardiac disorders) | 2/353 | 1/350
Angina pectoris (Cardiac disorders) | 1/353 | 2/350
Arrhythmia (Cardiac disorders) | 1/353 | 0/350
Atrial fibrillation (Cardiac disorders) | 1/353 | 2/350
Cardiac failure (Cardiac disorders) | 1/353 | 1/350
Cardiac failure congestive (Cardiac disorders) | 0/353 | 1/350
Myocardial infarction (Cardiac disorders) | 1/353 | 1/350
Gingival bleeding (Gastrointestinal disorders) | 1/353 | 0/350
Gingival recession (Gastrointestinal disorders) | 1/353 | 0/350
Inguinal hernia (Gastrointestinal disorders) | 0/353 | 1/350
Periodontal disease (Gastrointestinal disorders) | 1/353 | 0/350
Chest pain (General disorders) | 2/353 | 2/350
Cellulitis (Infections and infestations) | 1/353 | 0/350
Road traffic accident (Injury, poisoning and procedural complications) | 1/353 | 0/350
Stent occlusion (Injury, poisoning and procedural complications) | 0/353 | 1/350
Tibia fracture (Injury, poisoning and procedural complications) | 1/353 | 0/350
Diabetes mellitus (Metabolism and nutrition disorders) | 1/353 | 1/350
Ketoacidosis (Metabolism and nutrition disorders) | 0/353 | 1/350
Back pain (Musculoskeletal and connective tissue disorders) | 1/353 | 1/350
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/353 | 1/350
Cerebrovascular accident (Nervous system disorders) | 2/353 | 0/350
Cervical root pain (Nervous system disorders) | 1/353 | 0/350
Complex partial seizures (Nervous system disorders) | 1/353 | 0/350
Syncope (Nervous system disorders) | 1/353 | 1/350
Menorrhagia (Reproductive system and breast disorders) | 1/353 | 0/350
Testicular torsion (Reproductive system and breast disorders) | 1/353 | 0/350
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/353 | 0/350
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/353 | 0/350
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/353 | 0/350
Percutaneous coronary intervention (Surgical and medical procedures) | 0/353 | 1/350
Circulatory collapse (Vascular disorders) | 0/353 | 1/350
Intermittent claudication (Vascular disorders) | 0/353 | 1/350
Thrombosis (Vascular disorders) | 1/353 | 0/350
Angina unstable (Cardiac disorders) | 1/353 | 0/350
Cardiogenic shock (Cardiac disorders) | 0/353 | 1/350
Coronary artery disease (Cardiac disorders) | 1/353 | 0/350
Ventricular tachycardia (Cardiac disorders) | 0/353 | 1/350
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/353 | 1/350
Infected cyst (Infections and infestations) | 1/353 | 0/350
Infected skin ulcer (Infections and infestations) | 0/353 | 1/350
Pneumonia (Infections and infestations) | 0/353 | 1/350
Ankle fracture (Injury, poisoning and procedural complications) | 0/353 | 1/350
Hypovolaemia (Metabolism and nutrition disorders) | 0/353 | 1/350
Diabetic coma (Nervous system disorders) | 0/353 | 1/350
Renal failure acute (Renal and urinary disorders) | 0/353 | 1/350
Arteriosclerosis (Vascular disorders) | 1/353 | 0/350
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Varenicline (Var) | Placebo (Pbo)
Angina pectoris (Cardiac disorders) | 12/353 | 5/350
Abdominal distension (Gastrointestinal disorders) | 7/353 | 3/350
Abdominal pain upper (Gastrointestinal disorders) | 15/353 | 9/350
Constipation (Gastrointestinal disorders) | 23/353 | 7/350
Diarrhoea (Gastrointestinal disorders) | 22/353 | 18/350
Dry mouth (Gastrointestinal disorders) | 13/353 | 7/350
Dyspepsia (Gastrointestinal disorders) | 19/353 | 12/350
Flatulence (Gastrointestinal disorders) | 8/353 | 7/350
Nausea (Gastrointestinal disorders) | 104/353 | 30/350
Vomiting (Gastrointestinal disorders) | 29/353 | 4/350
Chest pain (General disorders) | 7/353 | 6/350
Fatigue (General disorders) | 25/353 | 14/350
Irritability (General disorders) | 6/353 | 9/350
Oedema peripheral (General disorders) | 7/353 | 4/350
Influenza (Infections and infestations) | 15/353 | 17/350
Nasopharyngitis (Infections and infestations) | 23/353 | 30/350
Upper respiratory tract infection (Infections and infestations) | 11/353 | 12/350
Back pain (Musculoskeletal and connective tissue disorders) | 13/353 | 8/350
Dizziness (Nervous system disorders) | 22/353 | 16/350
Dysgeusia (Nervous system disorders) | 16/353 | 8/350
Headache (Nervous system disorders) | 45/353 | 39/350
Somnolence (Nervous system disorders) | 2/353 | 7/350
Abnormal dreams (Psychiatric disorders) | 28/353 | 6/350
Anxiety (Psychiatric disorders) | 8/353 | 13/350
Insomnia (Psychiatric disorders) | 42/353 | 23/350
Nicotine dependence (Psychiatric disorders) | 9/353 | 5/350
Sleep disorder (Psychiatric disorders) | 12/353 | 5/350
Cough (Respiratory, thoracic and mediastinal disorders) | 7/353 | 13/350
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9/353 | 4/350
Hypertension (Vascular disorders) | 5/353 | 9/350

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 months (mo) from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.